CLINICAL TRIAL: NCT06735612
Title: Respiratory Syncytial Virus Infection in Exacerbations of Chronic Obstructive Pulmonary Diasease: the RECODE Study
Acronym: RECODE
Status: Recruiting | Type: Observational
Sponsor: Fundacio Privada Mon Clinic Barcelona (Other)
Responsible Party: Sponsor
Other Study IDs: RECODE
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Respiratory Synctial Virus; COPD; Chronic Obstructive Pulmonary Disease (COPD); Exacerbation of COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients during the RSV season
- Patients outside the RSV season

SUMMARY:
The goal of this observational study is to determine the prevalence of respiratory syncytial virus (RSV) infection and evaluate its association with clinical outcomes in patients with chronic obstructive pulmonary disease (COPD) who experience exacerbations during the RSV season (October-April). The main question it aims to answer is:

* What is the prevalence of RSV infection in patients with COPD during exacerbations in the RSV season?
* Does RSV infection lead to worse clinical outcomes, including hospitalization, longer length of stay, acute cardiovascular events, and/or death in patients with COPD exacerbations?

Researchers will compare patients with RSV infection to those without RSV infection to see if RSV infection results in worse clinical outcomes, such as increased hospitalization, longer stays, cardiovascular events, or death.

Participants will:

* Be adults diagnosed with COPD who present to the emergency department or day hospital due to acute exacerbations of their respiratory symptoms.
* Receive treatment as per standard clinical care for COPD exacerbations, including long-acting bronchodilators and inhaled corticosteroids, and may complete a course of antibiotics and/or oral corticosteroids if prescribed during hospitalization.
* Undergo diagnostic testing for RSV infection as part of the clinical routine to determine the presence or absence of the virus during their exacerbation.
* Have clinical outcomes monitored, including hospitalization rate, length of stay, and any acute cardiovascular events, as well as mortality during the exacerbation period.
* Provide relevant demographic and clinical data, including medical history, COPD severity, comorbidities, and previous exacerbation events.

ELIGIBILITY:
Inclusion Criteria:

* Female or male
* ≥50 years of age
* Seeking urgent medical attention because of ECOPD, as defined by the Rome consensus definition: "in a patient with COPD, an exacerbation is an event characterized by dyspnea and/or cough and sputum that worsen over <14 d, which may be accompanied by tachypnoea and/or tachycardia and is often associated with increased local and systemic inflammation caused by airway infection, pollution, or other insult to the airways"

Exclusion Criteria:

* Previous RSV vaccination (other vaccines will be allowed and recorded)
* Active cancer (or any other disease) that may alter the immune status of the patient
* Neurologic disorders that incapacitate the participation of the patient
* No signing of the informed consent

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with the presence of RSV infection (RSV+ considered as cases and RSV- considered as controls) in ECOPD at the Emergency Room or Day Hospital facilities.
Sampling Method: Non-Probability Sample
Enrollment: 892 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
To determine the prevalence of RSV infection because of ECOPD during the RSV season (October-April). | 1 year
  To determine the prevalence of RSV infection (defined as the detection of RSV by RT PCR in nasopharyngeal swab, saliva or sputum samples) among COPD patients seeking acute medical attention in the Emergency Room or Day Hospital facilities because of ECOPD during the RSV season (October-April).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínic de Barcelona, Barcelona, Spain